CLINICAL TRIAL: NCT03583099
Title: The CAPTURE Study: Validating a Unique Chronic Obstructive Pulmonary Disease (COPD) Case Finding Tool in Primary Care
Brief Title: The CAPTURE Study: Validating a Unique COPD Case Finding Tool in Primary Care (Aim 3)
Acronym: CAPTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Michigan (Other); National Jewish Health (Other); Wake Forest University Health Sciences (Other); Duke University (Other); High Plains Research Network (Network); L.A. Net Community Health Resource Network (Other); Oregon Health and Science University (Other); University of Kentucky (Other); University of Minnesota (Other); COPD Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1803019032-3; R01HL136682-01 (NIH)
Record Dates: First submitted 2018-03-05; First posted 2018-07-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participating primary practices will be randomized to one of 2 arms.
  * Arm 1: Practice clinicians will receive basic COPD education, and patient-level CAPTURE information with CAPTURE interpretation education (CAPTURE+ COPD education).
  * Arm 2: Practice clinicians will receive basic COPD education only (COPD education).
Who Masked: Participant, Care Provider
Masking Description: Practitioners at sites randomized to the COPD education only intervention will be blinded to CAPTURE scores.
  Practitioners in both intervention arms will be blinded to research spirometry results.
  Participants will be blinded to spirometry results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD Education (Active Comparator): Practice clinicians will receive basic COPD education only.
  Interventions: Other: COPD Education Only
- CAPTURE + COPD Education (Experimental): Practice clinicians will receive basic COPD education, and patient-level CAPTURE information with CAPTURE interpretation education. As the second aim address the optimal format for delivering practice CAPTURE education this will be incorporated at the sites randomized to this arm.
  Interventions: Other: COPD plus CAPTURE education and patient-level information

INTERVENTIONS:
Other: COPD plus CAPTURE education and patient-level information — Basic COPD Education plus CAPTURE education and patient-level CAPTURE information will be provided to all practice personnel randomized to the 'CAPTURE + COPD Education' arm.
  Arms: CAPTURE + COPD Education
Other: COPD Education Only — Practice clinicians will receive basic COPD education only. Patient-level CAPTURE information will not be provided.
  Arms: COPD Education

SUMMARY:
A prospective, multicenter study including a cross-section validation to define sensitivity and specificity of CAPTURE to identify previously undiagnosed patients with clinically significant Chronic Obstructive Pulmonary Disease (COPD), and its impact on clinical care across a broad range of primary care settings in a cluster randomized controlled clinical trial.

DETAILED DESCRIPTION:
This is a large prospective, multi-center study explore the impact of the CAPTURE tool on clinical care and patient outcomes across a broad range of primary care settings in a cluster randomized controlled clinical trial.

The CAPTURE tool consists of a 5-item self-administered questionnaire and selected use of peak expiratory flow (PEF) measurement, designed to identify clinically significant COPD.

The CAPTURE study will enroll approximately 5,000 patients across 100 participating primary care clinics associated with practice-based research networks (PBRNs). Participants will be assessed with the CAPTURE Tool and have research spirometry testing.

Participating primary care practices will be randomized in a 1:1 fashion to one of the following interventions:

* Arm 1: Practice clinicians will receive basic COPD education, and patient-level CAPTURE information with CAPTURE interpretation education (CAPTURE+ COPD education).
* Arm 2: Practice clinicians will receive basic COPD education only (COPD education) and will be blinded to patient-level CAPTURE information.

A predefined subgroup of participants will undergo longitudinal follow-up at 12 months to determine the impact of the CAPTURE Tool on clinical care and patient outcomes. Participant reported data will be collected through in-person visits, telephone and mail-based methodologies, depending upon practice site preferences and feasibility. Clinic site data will also be collected from the medical record to assess for changes in practice-level care.

Primary outcome measure changes have been made in this ClinicalTrials.gov record because a planned part of the primary outcome measure was inadvertently missing from the initial draft of the protocol. It has been added to this ClinicalTrials.gov record to align with the most recent IRB-approved protocol. Secondary outcome measure changes were initiated as driven by the literature and advances in accepted methods of management and categorization of patients with COPD. An additional secondary outcome measure was added due to the COVID-19 pandemic. The changes have been made in ClinicalTrials.gov to align with the most recent IRB-approved protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of signed and dated informed consent form
* 2. Stated willingness to comply with all study procedures and availability for the duration of the study
* 3. Male or female, aged 45 - 80 years
* 4. Able to read and speak English or Spanish

Exclusion Criteria:

* 1. Previous clinician provided diagnosis of COPD
* 2. Treated respiratory infection (with antibiotics and/or systemic steroids) in the past 30 days
* 3. Participants unable to perform spirometry due to any of the following conditions within the past 30 days

  1. Chest surgery
  2. Abdominal surgery
  3. Eye surgery
  4. Heart attack
  5. Stroke

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, MS, Principal Investigator — Weill Medical College of Cornell University; MeiLan Han, MD, MS, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - LANet, Los Angeles, California
  - High Plains Research Network, Aurora, Colorado
  - COPD Foundation, Miami, Florida
  - Cook County Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Circuit Clinical, Buffalo, New York
  - Atrium Healthcare, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Oregon Rural Practice-based Research Network (ORPRN), Portland, Oregon

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Practices
Groups:
- Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results: Practice clinicians received basic COPD education, CAPTURE education, and clinician receipt of patient-level CAPTURE screening results.
- Enhanced Usual Care: COPD Education: Practice clinicians received COPD education only.
Period: Overall Study
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Started | 1118; 51 Practices | 886; 48 Practices (One practice did not have any participants meeting the criteria for 12 month follow-up.)
Primary Analysis Population | 226; 49 Practices | 161; 44 Practices
Completed | 802; 51 Practices | 613; 46 Practices (Two practices did not have any participants meeting the criteria for 12 month follow-up.)
Not Completed | 316; 0 Practices | 273; 2 Practices

BASELINE CHARACTERISTICS:
Population: Participants with a spirometry consistent with obstruction (FEV1/FVC < 0.70); spirometry FEV1 <80% predicted, as well as a 5% random sample of all other participants underwent longitudinal follow-up at 12-months.
Units Other Than Participants: practices
Groups:
- Intervention Arm: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results: Intervention Arm: Practice clinicians received basic COPD education, CAPTURE education, and clinician receipt of patient-level CAPTURE screening results.
- Enhanced Usual Care Arm: COPD Education: Enhanced Usual Care Arm: Practice clinicians received basic COPD education only.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education | Total
Number analyzed (Participants) | 1118 | 886 | 2004
Number analyzed (practices) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62 (9) | 63 (9) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 677 | 530 | 1207
  Male | 441 | 356 | 797
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic/Non-Latino | 984 | 711 | 1695
  Hispanic or Latino | 89 | 149 | 238
  Don't Know/Prefer not to answer | 45 | 22 | 67
  Missing Data | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 362 | 236 | 598
  White | 642 | 514 | 1156
  Other than White or Black/African American | 62 | 44 | 106
  Don't know/Prefer not to answer | 52 | 90 | 142
  Missing Data | 0 | 2 | 2
Body Max Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 33 (8) | 33 (8) | 33 (8)
Enrollment Date [Count of Participants; unit: Participants]
  Before March 20, 2019 | 284 | 80 | 364
  March 20, 2019 - November 19, 2019 | 277 | 301 | 578
  Sep 20, 2019 - Mar 19, 2020 | 264 | 307 | 571
  Mar 20, 2020 or later | 293 | 198 | 491
Education [Count of Participants; unit: Participants]
  Less than high school | 128 | 118 | 246
  High school or GED | 298 | 231 | 529
  Vocational school or some college | 310 | 197 | 507
  College degree | 250 | 218 | 468
  Professional or graduate degree | 127 | 118 | 245
  Missing Data | 5 | 4 | 9
Employment [Count of Participants; unit: Participants]
  Working part-time or full-time | 198 | 141 | 339
  Not working for reason other than disability | 488 | 368 | 856
  Not working due to disability | 427 | 376 | 803
  Missing | 5 | 1 | 6
Health insurance [Count of Participants; unit: Participants]
  Private or both private and public insurance | 562 | 467 | 1029
  Public insurance or no insurance | 532 | 407 | 939
  Other/Don't know | 24 | 12 | 36
Participants with a history of asthma [Count of Participants; unit: Participants]
  True | 913 | 723 | 1636
  False | 203 | 162 | 365
  Missing | 2 | 1 | 3
Asthma and respiratory medication [Count of Participants; unit: Participants]
  No asthma, and no respiratory medication | 825 | 661 | 1486
  No asthma, but short-acting bronchodilator (SABD) or maintenance respiratory medication | 87 | 62 | 149
  No asthma with no respiratory medication | 67 | 45 | 112
  Asthma with SABD only | 59 | 54 | 113
  Asthma with maintenance respiratory medication | 77 | 62 | 139
  Missing Data | 3 | 2 | 5
Cigarette smoking [Count of Participants; unit: Participants]
  Never | 518 | 456 | 974
  Former | 373 | 283 | 656
  Current | 223 | 146 | 369
  Missing | 4 | 1 | 5
Maintenance respiratory medication [Count of Participants; unit: Participants]
  None | 1014 | 798 | 1812
  Inhaled Corticosteroids (ICS) alone | 31 | 22 | 53
  Long-acting brochodilator (LABA) and ICS | 63 | 55 | 118
  Other combination of LABA, Long-acting beta2-agonist (LAMA), and ICS | 9 | 10 | 19
  Missing Data | 1 | 1 | 2
Short-acting bronchodilator Use [Count of Participants; unit: Participants]
  True | 197 | 154 | 351
  False | 920 | 731 | 1651
  Missing Data | 1 | 1 | 2
Number of participants with a COPD Assessment Test (CAT) Score ≥ 10 [Count of Participants; unit: Participants] — The COPD Assessment Test is an 8-item self-administered questionnaire with scores ranging from 0 to 40. Scores ≥ 10 considered to represent significant respiratory symptom burden.
  Participants
    CAT score < 10 | 517 | 451 | 968
    CAT score ≥ 10 | 600 | 435 | 1035
    Missing Data | 1 | 0 | 1
Number of participants with Modified Medical Research Council dyspnea score ≥ 2 [Count of Participants; unit: Participants] — The Modified Medical Research Council Dyspnea Scale is used to assess the degree of baseline functional disability due to dyspnea. Scores range from 0 - 4. A higher the score indicates more dyspnea.
  Participants
    True | 831 | 682 | 1513
    False | 285 | 202 | 487
    Missing | 2 | 2 | 4
Acute respiratory illness in the past 12 months before baseline [Count of Participants; unit: Participants] — Queried as 'Over the last 12 months, have you had episodes of chest troubles (cough, phlegm, or shortness of breath) requiring treatment with antibiotics and/or steroids?'
  Participants
    True | 151 | 121 | 272
    False | 966 | 763 | 1729
    Missing | 1 | 2 | 3
Forced Vital Capacity (FVC) percent of predicted value [Mean (Standard Deviation); unit: percent predicted] — Post-bronchodilator for patients who completed post-bronchodilator spirometry; otherwise, pre-bronchodilator Population: Missing data from 16 participants in the Enhanced Usual Care Arm: COPD Education.
  Missing data from 31 participants in the Intervention Arm: COPD education plus CAPTURE education and patient-level CAPTURE screening results.
  percent predicted
    number analyzed (Participants) | 1087 | 870 | 1957
    (all) | 82 (16) | 84 (18) | 83 (17)
Forced Expiratory Volume in 1 second (FEV1), percent of predicted value [Mean (Standard Deviation); unit: percent predicted] — Post-bronchodilator for patients who completed post-bronchodilator spirometry; otherwise, pre-bronchodilator Population: Missing data from 16 participants in the Enhance Usual Care Arm: COPD education.
  Missing data from 31 participants in the Intervention Arm: COPD education plus CAPTURE education and patient-level CAPTURE screening results.
  percent predicted
    number analyzed (Participants) | 1087 | 870 | 1957
    (all) | 81 (16) | 82 (19) | 81 (17)
Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) mean [Mean (Standard Deviation); unit: percent] — Post-bronchodilator for patients who completed post-bronchodilator spirometry; otherwise, pre-bronchodilator Population: Missing data from 16 participants in the Enhanced Usual Care Arm: COPD Education Missing data from 31 participants in the Intervention Arm: COPD Education plus CAPTURE education and patient-level CAPTURE screening results
  percent
    number analyzed (Participants) | 1087 | 870 | 1957
    (all) | 77 (8) | 76 (8) | 76 (8)
Spirometry classification [Count of Participants; unit: Participants] — Normal Spirometry = COPD absent and FEV1 ≥ 80% predicted, Preserved ratio, impaired spirometry (PRISM) = COPD absent and FEV1 < 80% predicted
  Participants
    Normal spirometry | 478 | 382 | 860
    Preserved ratio, impaired spirometry | 372 | 278 | 650
    Spirometry-defined COPD | 180 | 164 | 344
    Undetermined | 88 | 62 | 150
CAPTURE question 5 response [Count of Participants; unit: Participants] — CAPTURE Question #5: In the past 12 months, how many times did you miss work, school, or other activities due to a cold, bronchitis, or pneumonia?
  Participants
    None | 810 | 672 | 1482
    Once | 154 | 109 | 263
    Two or more | 154 | 105 | 259
Practice Baseline Characteristic: Practice Type [Number; unit: practices]
  Part of large health system, Accountable Care Organization (ACO), or similar | 17 | 18 | 35
  Part of academic medical center/health system | 15 | 13 | 28
  Federally Qualified Health Center | 10 | 8 | 18
  Independent practice | 6 | 3 | 9
  Other | 2 | 5 | 7
  Missing | 1 | 1 | 2
Practice Baseline Characteristic: Number of primary care clinicians [Number; unit: practices] — Clinicians include physicians (MD or DO), nurse practitioners, and physician assistants.
  practices
    0 - 4 | 17 | 17 | 34
    5 -0 | 21 | 15 | 36
    10 or more | 11 | 14 | 25
    Missing | 2 | 2 | 4
Practice Baseline Characteristic: Practice is a residency site [Number; unit: practices]
  Yes | 13 | 7 | 20
  No | 37 | 40 | 77
  Missing | 1 | 1 | 2
Practice Baseline Characteristic: Spirometry is performed in-house [Number; unit: practices]
  Yes | 28 | 30 | 58
  No | 22 | 17 | 39
  Missing | 1 | 1 | 2
Practice Baseline Characteristic: Rural location [Number; unit: practices] — Practice is located in a ZIP code designated as rural by the Federal Office of Rural Health Policy.
  practices
    Yes | 10 | 8 | 18
    No | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Proportion of CAPTURE+ Participants Who Meet a Composite Endpoint for Diagnosis and Management of COPD
Description: Proportion of CAPTURE+ participants who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results: Intervention Arm: Practice clinicians received basic COPD education, CAPTURE education, and clinician receipt of patient-level CAPTURE screening results.
- Enhanced Usual Care: COPD Education: Enhanced Usual Care Arm: Practice clinicians received basic COPD education only.
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 45.9 [38.3 to 53.6] | 41.9 [34.0 to 49.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.47, generalized estimating equation contrast; Difference in proportion = 4.0, 95% CI 2-sided [-6.9 to 15.0] — The direction of the difference is Intervention: COPD education plus CAPTURE education and patient-level CAPTURE screening results minus the Enhanced Usual Care: COPD education

2. Secondary Outcome: Proportion of CAPTURE+ Participants Who Are Referred for or Complete Clinical Spirometry Testing
Description: CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: Participants who completed the 12-month follow-up survey, which required them to survive, were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 30.0 [22.2 to 37.9] | 19.6 [13.0 to 26.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.05, Generalized estimating equation contrast; Difference in proportion = 10.4, 95% CI 2-sided [0.1 to 20.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of CAPTURE+ Participants Who Are Newly Diagnosed With COPD
Description: CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Enhanced Usual Care Arm: COPD Education: Practice clinicians received basic COPD education only.
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 13.7 [8.6 to 18.7] | 12.4 [6.2 to 18.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.75, Generalized estimating equation contrast; Difference in proportion = 1.3, 95% CI 2-sided [-6.7 to 9.2] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of CAPTURE+ Participants With Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Enhanced Usual Care: COPD Education: Practice clinicians received basic COPD education only.
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 25.2 [19.2 to 31.2] | 27.9 [21.5 to 34.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.54, Generalized estimating equation contrast; Difference in proportion = -2.7, 95% CI 2-sided [-11.5 to 6.1] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Proportion of CAPTURE+ Participants Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 2
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 17.4 [11.8 to 23.1] | 12.3 [7.8 to 16.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.16, Generalized estimating equation contrast; Difference in proportion = 5.1, 95% CI 2-sided [-2.1 to 12.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Proportion of CAPTURE+ Participants Who Are Referred for or Complete Pulmonary Rehabilitation
Description: as for outcome 2
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 6.40 [2.40 to 10.3] | 7.00 [2.90 to 11.20]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.82, Generalized estimating equation contrast; Difference in proportion = -0.6, 95% CI 2-sided [-6.4 to 5.1] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Proportion of CAPTURE+ Participants Who Have Received a Recommendation for, or Administration of Influenza Vaccination.
Description: as for outcome 2
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 84.5 [79.4 to 89.5] | 90.8 [86.4 to 95.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.06, Generalized estimating equation contrast; Difference in proportion = -6.3, 95% CI 2-sided [-13.0 to 0.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Proportion of CAPTURE+ Participants Smoking at the Baseline With Any Components of the Primary Endpoint OR Any of the 4 Events Described in the Description Below.
Description: Proportion of CAPTURE+ participants currently smoking at the baseline visit who have any of the components of the Aim 3 primary endpoint: 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  OR
  1) clinical counseling or recommendation for smoking cessation, 2) referral to a smoking cessation program, 3) referral to a smoking quit line, 4) newly prescribed medication for smoking cessation.
  CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline who had complete follow-up data for all elements of the composite endpoints available were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 49 | 25
percent | 83.37 [82.70 to 84.03] | 85.90 [73.93 to 97.87]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.68, Generalized estimating equation contrast; Difference in proportion = -2.5, 95% CI 2-sided [-14.5 to 9.5] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Are Referred for or Complete Clinical Spirometry Testing
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 37.52 [24.67 to 50.37] | 24.19 [8.80 to 39.58]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.19, Generalized estimating equation contrast; Difference in proportion = 13.3, 95% CI 2-sided [-6.72 to 33.38] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive a New Diagnosis of COPD
Description: as for outcome 3
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 24.62 [13.48 to 35.78] | 23.77 [8.80 to 38.74]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.93, Generalized estimating equation contrast; Difference in proportion = 0.85, 95% CI 2-sided [-17.82 to 19.52] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Are Newly Prescribed Respiratory Medication
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 37.05 [26.73 to 47.37] | 30.22 [15.88 to 44.57]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.45, Generalized estimating equation contrast; Difference in proportion = 6.83, 95% CI 2-sided [-10.84 to 24.50] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive a Referral to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 21.58 [9.55 to 33.62] | 13.98 [0.36 to 27.61]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.41, Generalized estimating equation contrast; Difference in proportion = 7.6, 95% CI 2-sided [-10.58 to 25.78] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive a Referral for, or Complete Pulmonary Rehabilitation.
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 12.01 [2.62 to 21.40] | 10.16 [-1.57 to 21.88]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.81, Generalized estimating equation contrast; Difference in proportion = 1.85, 95% CI 2-sided [-13.17 to 16.88] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive Clinician Counseling or Recommendation for Smoking Cessation
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 71.98 [58.59 to 85.36] | 63.96 [44.78 to 83.15]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.51, Generalized estimating equation contrast; Difference in proportion = 8.01, 95% CI 2-sided [-15.38 to 31.40] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive a Referral to a Smoking Cessation Program
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline who had follow-up data available for referral information for smoking cessation programs were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 50 | 25
percent | 30.36 [16.69 to 44.03] | 40.70 [20.46 to 60.95]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.41, Generalized estimating equation contrast; Difference in proportion = -10.34, 95% CI 2-sided [-34.78 to 14.09] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Proportion of CAPTURE+ Participants Capture Positive Participants Currently Smoking at Baseline Who Referral to a Smoking Quit Line
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline who had follow-up data available for referral information for a smoking quit line were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 49 | 25
percent | 55.60 [39.32 to 71.88] | 59.54 [37.88 to 81.19]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.76, Generalized estimating equation contrast; Difference in proportion = -3.94, 95% CI 2-sided [-31.03 to 23.16] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Receive a Newly Prescribed Medication for Smoking Cessation.
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants currently smoking at baseline who had follow-up data for newly prescribed medication for smoking cessation were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 49 | 25
percent | 55.14 [40.73 to 69.55] | 55.90 [35.97 to 75.83]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.95, Generalized estimating equation contrast; Difference in proportion = -0.76, 95% CI 2-sided [-25.36 to 23.83] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: 12-month Change in COPD Assessment Test (CAT) Score (12 Month CAT Change) in CAPTURE+ Participants
Description: The COPD Assessment Test (CAT) is scored 0-40. Higher score = more severe COPD impact.
  CAPTURE+ is defined as a CAPTURE score ≥ 5, or CAPTURE score 2, 3, or 4 with low PEF (<350 L/min for males,<250 L/min for females). Higher values = higher likelihood of COPD.
  The mixed model for 12 month CAT change was: 12 month CAT change = intercept (Enhanced Usual Care (EUC) parameter) + slope (difference between Intervention and EUC) + practice random intercept. 12 month change units are CAT score differences; ie. if 12 month CAT change = 1, CAT score increased by 1 point in 12 months.
  Intercept term estimates mean EUC 12 month CAT change. The intercept + slope terms estimate mean intervention group 12 month CAT change.
  The slope estimates mean 12 month CAT change differences between Intervention versus EUC where difference direction is: Intervention results minus the EUC results; ie. if the slope = 1, the intervention group had 1 point higher 12 month CAT change compared to EUC.
Time Frame: Baseline to 12 months
Population: There was missing data from 2 participants in the Enhanced Usual Care arm and missing data from 4 participants in the Intervention arm.
Measure: Mean (95% Confidence Interval); unit: CAT score point scale
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 222 | 159
CAT score point scale | -1.25 [-2.33 to -0.18] | -0.93 [-2.21 to 0.34]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.55, Mixed Models Analysis — The p-value is adjusted for baseline CAT score; Difference in means = -0.32, 95% CI 2-sided [-2.01 to 1.36] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Proportion of CAPTURE+ Participants Who Experience Exacerbations.
Description: CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
  Exacerbation is defined as acute respiratory illness requiring antibiotic/steroid during follow-up.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
percent | 23.9 [17.2 to 30.7] | 15.3 [9.7 to 20.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.05, Generalized estimating equation contrast; Difference in proportion = 8.7, 95% CI 2-sided [-0.1 to 17.4] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with clinically significant COPD who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation. (composite endpoint)
  Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 50.05 [33.83 to 66.27] | 48.25 [31.56 to 64.94]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.88, Generalized estimating equation contrast; Difference in proportion = 1.81, 95% CI 2-sided [-21.47 to 25.08] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Proportion of Participants With Clinically Significant COPD With a Referral for or Completion of Clinical Spirometry Testing
Description: Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 17.42 [5.72 to 29.13] | 23.04 [9.91 to 36.17]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.53, Generalized estimating equation contrast; Difference in proportion = -5.62, 95% CI 2-sided [-23.21 to 11.97] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Proportion of Participants With Clinically Significant COPD With a New Diagnosis of COPD
Description: Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 24.26 [10.39 to 38.12] | 13.58 [2.18 to 24.97]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.24, Generalized estimating equation contrast; Difference in proportion = 10.68, 95% CI 2-sided [-7.27 to 28.63] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Proportion of Participants With Clinically Significant COPD With a Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 24.87 [11.58 to 38.16] | 38.42 [23.34 to 53.50]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.19, Generalized estimating equation contrast; Difference in proportion = -13.55, 95% CI 2-sided [-33.65 to 6.55] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Proportion of Participants With Clinically Significant COPD With a Referral to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 10.14 [0.95 to 19.33] | 9.76 [0.72 to 18.80]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.95, Generalized estimating equation contrast; Difference in proportion = 0.38, 95% CI 2-sided [-12.50 to 13.27] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Proportion of Participants With Clinically Significant COPD With a Referral for or Completion of Pulmonary Rehabilitation.
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 5.63 [-0.79 to 12.06] | 12.61 [6.10 to 19.11]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.14, Generalized estimating equation contrast; Difference in proportion = -6.97, 95% CI 2-sided [-16.12 to 2.17] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Who Receive a Recommendation for or Administration of Influenza Vaccination
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for clinically significant COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 40 | 39
percent | 93.22 [84.33 to 102.11] | 94.28 [85.74 to 102.82]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.87, Generalized estimating equation contrast; Difference in proportion = -1.06, 95% CI 2-sided [-13.39 to 11.27] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Proportion of Participants With Spirometric COPD Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with spirometric COPD who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 34.5 [24.1 to 44.8] | 36.2 [26.6 to 45.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.81, Generalized estimating equation contrast; Difference in proportion = -1.8, 95% CI 2-sided [-15.9 to 12.4] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Proportion of Participants With Spirometric COPD Referred for or Completion of Clinical Spirometry Testing
Description: Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 17.4 [10.2 to 24.7] | 15.1 [9.1 to 21.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.63, Generalized estimating equation contrast; Difference in proportion = 2.3, 95% CI 2-sided [-7.2 to 11.8] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Proportion of Participants With Spirometric COPD With a New Diagnosis of COPD.
Description: Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 15.9 [9.4 to 22.4] | 10.1 [4.9 to 15.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.17, Generalized estimating equation contrast; Difference in proportion = 5.8, 95% CI 2-sided [-2.5 to 14.2] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Proportion of Participants With Spirometric COPD With Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 19.8 [12.1 to 27.5] | 22.7 [16.1 to 29.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.58, Generalized estimating equation contrast; Difference in proportion = -2.9, 95% CI 2-sided [-13.0 to 7.3] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Proportion of Participants With Spirometric COPD Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 7.6 [2.3 to 12.9] | 8.1 [2.5 to 13.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.89, Generalized estimating equation contrast; Difference in proportion = -0.6, 95% CI 2-sided [-8.3 to 7.1] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Proportion of Participants With Spirometric COPD Who Are Referred for or Complete Pulmonary Rehabilitation.
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 4.0 [0.7 to 7.2] | 7.8 [3.6 to 12.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.16, Generalized estimating equation contrast; Difference in proportion = -3.9, 95% CI 2-sided [-9.2 to 1.5] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Proportion of Participants With Spirometric COPD Who Receive a Recommendation for or Administration of Influenza Vaccination.
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for spirometric COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 126 | 119
percent | 87.6 [81.4 to 93.7] | 89.8 [83.6 to 95.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.62, Generalized estimating equation contrast; Difference in proportion = -2.2, 95% CI 2-sided [-10.9 to 6.5] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Proportion of Participants With Mild COPD Who Meet Any of the Components of the Primary Endpoint
Description: Proportion of participants with Mild COPD who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7 plus both of the following: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 27.02 [16.48 to 37.57] | 28.66 [17.13 to 40.20]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.84, Generalized estimating equation contrast; Difference in proportion = -1.64, 95% CI 2-sided [-17.27 to 13.99] — [estimate comment as in outcome 1, analysis 1]

35. Secondary Outcome: Proportion of Participants With Mild COPD Referred for or Completion of Clinical Spirometry Testing
Description: Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7 plus both of the following: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 17.25 [9.16 to 25.34] | 11.16 [4.13 to 18.20]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.27, Generalized estimating equation contrast; Difference in proportion = 6.09, 95% CI 2-sided [-4.63 to 16.80] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Proportion of Participants With Mild COPD With a New Diagnosis of COPD
Description: Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7 plus both of the following: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 11.36 [4.38 to 18.34] | 8.45 [2.00 to 14.89]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.55, Generalized estimating equation contrast; Difference in proportion = 2.91, 95% CI 2-sided [-6.59 to 12.41] — [estimate comment as in outcome 1, analysis 1]

37. Secondary Outcome: Proportion of Participants With Mild COPD With a Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7 plus both of the following: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 17.29 [9.13 to 25.45] | 14.92 [6.87 to 22.97]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.69, Generalized estimating equation contrast; Difference in proportion = 2.37, 95% CI 2-sided [-9.09 to 13.83] — [estimate comment as in outcome 1, analysis 1]

38. Secondary Outcome: Proportion of Participants With Mild COPD Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 5.89 [0.03 to 11.74] | 5.53 [-0.62 to 11.68]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.93, Generalized estimating equation contrast; Difference in proportion = 0.36, 95% CI 2-sided [-8.13 to 8.85] — [estimate comment as in outcome 1, analysis 1]

39. Secondary Outcome: Proportion of Participants With Mild COPD Referred for or Completion of Pulmonary Rehabilitation.
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 3.49 [-0.39 to 7.37] | 7.50 [1.72 to 13.27]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.26, Generalized estimating equation contrast; Difference in proportion = -4.01, 95% CI 2-sided [-10.97 to 2.95] — [estimate comment as in outcome 1, analysis 1]

40. Secondary Outcome: Proportion of Participants With Mild COPD Who Received a Recommendation or Administration of Influenza Vaccination.
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 86 | 80
percent | 85.04 [76.43 to 93.64] | 87.07 [78.36 to 95.79]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.74, Generalized estimating equation contrast; Difference in proportion = -2.04, 95% CI 2-sided [-14.28 to 10.21] — [estimate comment as in outcome 1, analysis 1]

41. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with preserved ratio, impaired spirometry (PRISm) who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 30.4 [25.2 to 35.7] | 30.4 [24.3 to 36.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.98, Generalized estimating equation contrast; Difference in proportion = 0.1, 95% CI 2-sided [-7.9 to 8.1] — [estimate comment as in outcome 1, analysis 1]

42. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Referred for or Completion of Clinical Spirometry Testing.
Description: Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 18.5 [14.1 to 22.9] | 15.9 [10.5 to 21.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.46, Generalized estimating equation contrast; Difference in proportion = 2.6, 95% CI 2-sided [-4.3 to 9.6] — [estimate comment as in outcome 1, analysis 1]

43. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) With New Diagnosis of COPD.
Description: Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 7.4 [4.3 to 10.5] | 5.8 [2.5 to 9.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.50, Generalized estimating equation contrast; Difference in proportion = 1.5, 95% CI 2-sided [-3.0 to 6.1] — [estimate comment as in outcome 1, analysis 1]

44. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) With a Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 17.4 [12.9 to 21.9] | 17.5 [12.6 to 22.5]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.96, Generalized estimating equation contrast; Difference in proportion = -0.2, 95% CI 2-sided [-6.8 to 6.5] — [estimate comment as in outcome 1, analysis 1]

45. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 13.4 [9.8 to 17.1] | 11.2 [7.5 to 14.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.40, Generalized estimating equation contrast; Difference in proportion = 2.2, 95% CI 2-sided [-3.0 to 7.5] — [estimate comment as in outcome 1, analysis 1]

46. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Referred for or Completion of Pulmonary Rehabilitation.
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 4.4 [1.9 to 7.0] | 4.6 [1.3 to 7.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.96, Generalized estimating equation contrast; Difference in proportion = -0.1, 95% CI 2-sided [-4.3 to 4.0] — [estimate comment as in outcome 1, analysis 1]

47. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Who Receive a Recommendation for or Administration of Influenza Vaccination.
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for preserved ratio, impaired spirometry (PRISm) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 271 | 189
percent | 85.2 [80.2 to 90.2] | 85.1 [78.9 to 91.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.98, Generalized estimating equation contrast; Difference in proportion = 0.1, 95% CI 2-sided [-7.9 to 8.1] — [estimate comment as in outcome 1, analysis 1]

48. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with symptomatic non-obstructed (SNO) meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC<0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10. The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 28.4 [21.6 to 35.2] | 32.6 [23.9 to 41.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.46, Generalized estimating equation contrast; Difference in proportion = -4.2, 95% CI 2-sided [-15.2 to 6.8] — [estimate comment as in outcome 1, analysis 1]

49. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Referred for or Completion of Clinical Spirometry Testing.
Description: Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC < 0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10.
  The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 18.8 [13.1 to 24.5] | 14.9 [8.6 to 21.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.37, Generalized estimating equation contrast; Difference in proportion = 3.9, 95% CI 2-sided [-4.7 to 12.4] — [estimate comment as in outcome 1, analysis 1]

50. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) With a New Diagnosis of COPD
Description: Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC < 0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10.
  The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
  A new diagnosis of COPD is defined as COPD recorded in the participant's chart or reported by the participant via the follow-up survey.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 4.8 [1.5 to 8.2] | 5.7 [1.7 to 9.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.75, Generalized estimating equation contrast; Difference in proportion = -0.8, 95% CI 2-sided [-6.0 to 4.4] — [estimate comment as in outcome 1, analysis 1]

51. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC < 0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10.
  The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 12.3 [7.1 to 17.5] | 21.0 [13.0 to 29.1]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.08, Generalized estimating equation contrast; Difference in proportion = -8.7, 95% CI 2-sided [-18.3 to 0.9] — [estimate comment as in outcome 1, analysis 1]

52. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 6.0 [2.8 to 9.2] | 10.8 [5.9 to 15.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.11, Generalized estimating equation contrast; Difference in proportion = -4.8, 95% CI 2-sided [-10.6 to 1.1] — [estimate comment as in outcome 1, analysis 1]

53. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Referred for or Completion of Pulmonary Rehabilitation.
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 5.4 [1.6 to 9.3] | 5.0 [1.1 to 9.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.89, Generalized estimating equation contrast; Difference in proportion = 0.4, 95% CI 2-sided [-5.1 to 5.9] — [estimate comment as in outcome 1, analysis 1]

54. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Who Receive a Recommendation or Administration of Influenza Vaccination.
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 186 | 127
percent | 80.4 [73.9 to 86.8] | 89.1 [83.2 to 95.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.05, Generalized estimating equation contrast; Difference in proportion = -8.8, 95% CI 2-sided [-17.5 to -0.0] — [estimate comment as in outcome 1, analysis 1]

55. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of CAPTURE+ participants enrolled before March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 52.81 [41.97 to 63.65] | 36.04 [19.64 to 52.44]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.09, Generalized estimating equation contrast; Difference in proportion = 16.76, 95% CI 2-sided [-2.89 to 36.42] — [estimate comment as in outcome 1, analysis 1]

56. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of CAPTURE+ participants enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 45.7 [36.9 to 54.5] | 42.0 [33.5 to 50.5]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.56, Generalized estimating equation contrast; Difference in proportion = 3.7, 95% CI 2-sided [-8.6 to 15.9] — [estimate comment as in outcome 1, analysis 1]

57. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Are Referred for or Complete Clinical Spirometry Testing
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 28.86 [13.70 to 44.02] | 18.45 [-7.20 to 44.10]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.49, Generalized estimating equation contrast; Difference in proportion = 10.41, 95% CI 2-sided [-19.39 to 40.20] — [estimate comment as in outcome 1, analysis 1]

58. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Are Referred for or Complete Clinical Spirometry Testing
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 30.4 [21.2 to 39.5] | 19.6 [12.8 to 26.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.06, Generalized estimating equation contrast; Difference in proportion = 10.8, 95% CI 2-sided [-0.5 to 22.1] — [estimate comment as in outcome 1, analysis 1]

59. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Are Newly Diagnosed With COPD
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 13.11 [6.46 to 19.75] | 12.70 [3.46 to 21.93]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.94, Generalized estimating equation contrast; Difference in proportion = 0.41, 95% CI 2-sided [-10.97 to 11.79] — [estimate comment as in outcome 1, analysis 1]

60. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Are Newly Diagnosed With COPD
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 14.8 [8.5 to 21.1] | 12.1 [5.4 to 18.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.57, Generalized estimating equation contrast; Difference in proportion = 2.7, 95% CI 2-sided [-6.5 to 11.8] — [estimate comment as in outcome 1, analysis 1]

61. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 With Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low PEF, defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 24.15 [14.09 to 34.21] | 22.79 [6.23 to 39.34]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.89, Generalized estimating equation contrast; Difference in proportion = 1.36, 95% CI 2-sided [-18.01 to 20.73] — [estimate comment as in outcome 1, analysis 1]

62. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 With Newly Prescribed Respiratory Medication
Description: as for outcome 61
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 26.1 [19.2 to 33.0] | 28.4 [21.4 to 35.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.65, Generalized estimating equation contrast; Difference in proportion = -2.2, 95% CI 2-sided [-12.1 to 7.6] — [estimate comment as in outcome 1, analysis 1]

63. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 19.78 [8.65 to 30.91] | 7.30 [-6.18 to 20.77]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.16, Generalized estimating equation contrast; Difference in proportion = 12.48, 95% CI 2-sided [-5.00 to 29.96] — [estimate comment as in outcome 1, analysis 1]

64. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 16.9 [10.5 to 23.4] | 12.7 [8.1 to 17.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.29, Generalized estimating equation contrast; Difference in proportion = 4.3, 95% CI 2-sided [-3.6 to 12.2] — [estimate comment as in outcome 1, analysis 1]

65. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Are Referred for or Complete Pulmonary Rehabilitation
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 11.34 [3.31 to 19.37] | 6.06 [-4.60 to 16.72]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.44, Generalized estimating equation contrast; Difference in proportion = 5.28, 95% CI 2-sided [-8.07 to 18.62] — [estimate comment as in outcome 1, analysis 1]

66. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Are Referred for or Complete Pulmonary Rehabilitation
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 5.2 [1.0 to 9.4] | 6.8 [2.4 to 11.1]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.62, Generalized estimating equation contrast; Difference in proportion = -1.5, 95% CI 2-sided [-7.6 to 4.5] — [estimate comment as in outcome 1, analysis 1]

67. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Have Received a Recommendation for, or Administration of Influenza Vaccination
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 88.30 [78.14 to 98.46] | 95.39 [82.91 to 108.87]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.39, Generalized estimating equation contrast; Difference in proportion = -7.1, 95% CI 2-sided [-23.18 to 9.0] — [estimate comment as in outcome 1, analysis 1]

68. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Have Received a Recommendation for, or Administration of Influenza Vaccination
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 83.3 [77.7 to 89.0] | 89.9 [85.2 to 94.5]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.08, Generalized estimating equation contrast; Difference in proportion = -6.6, 95% CI 2-sided [-13.9 to 0.8] — [estimate comment as in outcome 1, analysis 1]

69. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Have Received a Recommendation for, or Administration of Influenza Vaccination
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 53 | 29
percent | 71.66 [59.76 to 83.57] | 82.70 [69.16 to 96.24]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.23, Generalized estimating equation contrast; Difference in proportion = -11.30, 95% CI 2-sided [-29.06 to 7.00] — [estimate comment as in outcome 1, analysis 1]

70. Secondary Outcome: 12-month Change in COPD Assessment Test (CAT) Score (12 Month CAT Change) in CAPTURE+ Participants Enrolled Before March 20, 2019
Description: as for outcome 18
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Mean (95% Confidence Interval); unit: CAT score point scale
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
CAT score point scale | -2.44 [-5.08 to 0.20] | -1.30 [-6.50 to 3.90]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.97, Generalized estimating equation contrast — The p-value adjusts for baseline CAT score; Difference in means = -1.14, 95% CI 2-sided [-6.42 to 4.13] — [estimate comment as in outcome 1, analysis 1]

71. Secondary Outcome: 12-month Change in COPD Assessment Test (CAT) Score (12 Month CAT Change) in CAPTURE+ Participants Enrolled on or After March 20, 2019
Description: as for outcome 18
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Mean (95% Confidence Interval); unit: CAT score point scale
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
CAT score point scale | -0.92 [-2.15 to 0.31] | -0.92 [-2.28 to 0.44]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.47, Generalized estimating equation contrast; Difference in means = -0.003, 95% CI 2-sided [-1.86 to 1.85] — [estimate comment as in outcome 1, analysis 1]

72. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Experience Exacerbations.
Description: CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low peak expiratory flow (PEF), defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
  Exacerbation is defined as acute respiratory illness requiring antibiotic/steroid during follow-up.
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 26.62 [16.12 to 37.13] | 8.78 [-2.61 to 20.18]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.02, Generalized estimating equation contrast; Difference in proportion = 17.84, 95% CI 2-sided [2.34 to 33.34] — [estimate comment as in outcome 1, analysis 1]

73. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Experience Exacerbations.
Description: CAPTURE+ is defined as Participants with: CAPTURE score ≥ 5, or CAPTURE score of 2, 3, or 4 with a low peak expiratory flow (PEF), defined as <350 L/min for males and <250 L/min for females.
  CAPTURE scores range from 0 to 6. Higher values represent a higher likelihood of having clinically significant COPD.
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 23.7 [15.8 to 31.6] | 15.9 [10.0 to 21.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.12, Generalized estimating equation contrast; Difference in proportion = 7.8, 95% CI 2-sided [-2.0 to 17.6] — [estimate comment as in outcome 1, analysis 1]

74. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 Who Meet Any of Components of the Primary Endpoints.
Description: Proportion of participants with clinically significant COPD enrolled before March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 42.8 [6.20 to 79.5] | 0 [NA to NA] — Only one participant was in the Enhanced Usual Care group (insufficient data for confidence limits)
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 1.0, Fisher Exact; The p-value is calculated from a two-sided Fisher's exact test. This test is appropriate since only one outcome per practice was seen

75. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 Who Meet Any of Components of the Primary Endpoints.
Description: Proportion of participants with clinically significant COPD enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Clinically significant COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7, plus one of the following: 1) FEV1 < 60% predicted or > 1 exacerbation like event within the past 12 months.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 51.76 [33.74 to 69.77] | 49.69 [32.76 to 66.63]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.87, Generalized estimating equation contrast; Difference in proportion = 2.06, 95% CI 2-sided [-22.67 to 26.79] — [estimate comment as in outcome 1, analysis 1]

76. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 With a Referral for or Completion of Clinical Spirometry Testing
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for clinically significant COPD enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 14.3 [0 to 40.2] | 0 [NA to NA] — Only one participant was in the Enhanced Usual Care group (insufficient data for confidence limits)
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 1.0, Fisher Exact; The p-value is calculated from a two-sided Fisher's exact test

77. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 With a Referral for or Completion of Clinical Spirometry Testing
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for clinically significant COPD enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 18.14 [5.02 to 31.26] | 23.66 [10.19 to 37.14]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.56, Generalized estimating equation contrast; Difference in proportion = -5.53, 95% CI 2-sided [-24.33 to 13.28] — [estimate comment as in outcome 1, analysis 1]

78. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 With a New Diagnosis of COPD
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for clinically significant COPD enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 14.3 [0 to 40.2] | 0 [NA to NA] — Only one participant was in the Enhanced Usual Care group (insufficient data for confidence limits)
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 1.0, Fisher Exact; The p-value is calculated from a two-sided Fisher's exact test

79. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 a New Diagnosis of COPD
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 26.62 [10.75 to 42.49] | 13.96 [2.28 to 25.65]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.21, Generalized estimating equation contrast; Difference in proportion = 12.66, 95% CI 2-sided [-7.05 to 32.37] — [estimate comment as in outcome 1, analysis 1]

80. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 With a Newly Prescribed Respiratory Medication
Description: as for outcome 23
Time Frame: Baseline to 12 months
Population: as for outcome 78
Measure: Number (90% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 42.8 [6.20 to 79.5] | 0 [NA to NA] — Only one participant was in the Enhanced Usual Care group (insufficient data for confidence limits)
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 1.0, Fisher Exact; The p-value is calculated from a two-sided Fisher's exact test

81. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 With a Newly Prescribed Respiratory Medication
Description: as for outcome 23
Time Frame: Baseline to 12 months
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 21.04 [7.40 to 34.68] | 39.33 [24.21 to 54.45]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.08, Generalized estimating equation contrast; Difference in proportion = -18.29, 95% CI 2-sided [-38.66 to 2.08] — [estimate comment as in outcome 1, analysis 1]

82. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 With a Referral to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 14.3 [0 to 40.2] | 0 [NA to NA] — Only one participant was in the Enhanced Usual Care group (insufficient data for confidence limits)
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 1.0, Fisher Exact; The p-value is calculated from a two-sided Fisher's exact test

83. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 With a Referral to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 9.31 [-0.38 to 19.00] | 9.98 [0.75 to 19.21]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.92, Generalized estimating equation contrast; Difference in proportion = -0.67, 95% CI 2-sided [-14.06 to 12.71] — [estimate comment as in outcome 1, analysis 1]

84. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 With a Referral for or Completion of Pulmonary Rehabilitation
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program. | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program.

85. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled on or After March 20, 2019 With a Referral for or Completion of Pulmonary Rehabilitation
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 6.54 [-0.94 to 14.03] | 12.02 [5.03 to 19.01]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.29, Generalized estimating equation contrast; Difference in proportion = -5.47, 95% CI 2-sided [-15.72 to 4.77] — [estimate comment as in outcome 1, analysis 1]

86. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled Before March 20, 2019 Who Receive a Recommendation for or Administration of Influenza Vaccination (Abbreviated as Proportion in the Description)
Description: Clinically significant COPD = post-bronchodilator FEV1/FVC <0.7, plus: 1) FEV1 < 60% predicted or 2) > 1 exacerbation like event in the last year.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome.
  EUC proportion = intercept. Intervention proportion = intercept + slope.
  Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcomes between subjects in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 78
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 7 | 1
percent | 100 [NA to NA] — 100% (7 out of 7 participants) received recommendations for or administration of influenza vaccine. In this case, the raw number of 100% is reported without corresponding (unavailable) confidence limits. | 100 [NA to NA] — 100% (1 out of 1 participants) received recommendations for or administration of influenza vaccine. In this case, the raw number of 100% is reported without corresponding (unavailable) confidence limits.

87. Secondary Outcome: Proportion of Participants With Clinically Significant COPD Enrolled After August 13, 2020 Who Receive a Recommendation for or Administration of Influenza Vaccination
Description: as for outcome 21
Time Frame: Baseline to 12 months
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 33 | 38
percent | 91.13 [79.88 to 102.39] | 94.00 [85.24 to 102.77]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.69, Generalized estimating equation contrast; Difference in proportion = -2.87, 95% CI 2-sided [-17.14 to 11.39] — [estimate comment as in outcome 1, analysis 1]

88. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 Who Meet Any of the Components of the Primary Endpoint
Description: Proportion of participants with spirometric COPD enrolled before March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation
  Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for spirometric COPD enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | 16.03 [0.59 to 31.46] | 29.18 [8.37 to 49.98]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.32, Generalized estimating equation contrast; Difference in proportion = -13.15, 95% CI 2-sided [-39.06 to 12.76] — [estimate comment as in outcome 1, analysis 1]

89. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 Who Meet Any of the Components of the Primary Endpoint
Description: Proportion of participants with spirometric COPD enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation
  Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for spirometric COPD enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 37.0 [25.7 to 48.2] | 37.2 [27.0 to 47.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.98, Generalized estimating equation contrast; Difference in proportion = -0.2, 95% CI 2-sided [-15.5 to 15.0] — [estimate comment as in outcome 1, analysis 1]

90. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 Referred for or Completion of Clinical Spirometry Testing (Abbreviated as Proportion in the Description)
Description: Spirometric COPD: post-bronch FEV1/FVC <0.7. If only pre-bronch spirometry is available and FEV1/FVC < 0.65, subject will be considered to have COPD.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome.
  EUC proportion = intercept. Intervention proportion = intercept + slope.
  Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcomes between subjects in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | NA [NA to NA] — Only 1 of 17 subjects was referred for or completed spirometry testing (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of spirometric COPD subjects in practices and potential correlation of outcomes between individuals in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster. | 0 [NA to NA] — 0% (0 out of 8 participants) received referral for or completed of clinical spirometry testing. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits.

91. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 19.3 [11.3 to 27.2] | 16.2 [10.0 to 22.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.55, Generalized estimating equation contrast; Difference in proportion = 3.1, 95% CI 2-sided [-7.0 to 13.1] — [estimate comment as in outcome 1, analysis 1]

92. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 With a New Diagnosis of COPD
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | 5.10 [-4.64 to 14.64] | 13.71 [-5.55 to 32.96]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.43, Generalized estimating equation contrast; Difference in proportion = -8.61, 95% CI 2-sided [-30.19 to 12.97] — [estimate comment as in outcome 1, analysis 1]

93. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 With a New Diagnosis of COPD
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 17.5 [10.4 to 24.6] | 9.9 [4.4 to 15.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.10, Generalized estimating equation contrast; Difference in proportion = 7.6, 95% CI 2-sided [-1.4 to 16.5] — [estimate comment as in outcome 1, analysis 1]

94. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 With Newly Prescribed Respiratory Medication
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Spirometric COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC <0.7. If a participant is unable to complete a post-bronchodilator spirometry (refusal, technical error on the part of coordinator, etc.), and the pre-bronchodilator FEV1/FVC is less than 0.65, the participant will be considered to have COPD for the purpose of follow-up in this study.
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | 15.75 [0.71 to 30.79] | 14.93 [0.12 to 29.73]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.94, Generalized estimating equation contrast; Difference in proportion = 0.82, 95% CI 2-sided [-20.92 to 21.92] — [estimate comment as in outcome 1, analysis 1]

95. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 With Newly Prescribed Respiratory Medication
Description: as for outcome 94
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 20.1 [11.7 to 28.5] | 23.5 [16.4 to 30.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.55, Generalized estimating equation contrast; Difference in proportion = -3.4, 95% CI 2-sided [-14.4 to 7.6] — [estimate comment as in outcome 1, analysis 1]

96. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment (Abbreviated as Proportion in the Description)
Description: Spirometric COPD: post-bronch FEV1/FVC <0.7. If only pre-bronch spirometry is available and FEV1/FVC < 0.65, participant will be considered to have COPD.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome.
  EUC proportion = intercept. Intervention proportion = intercept + slope. Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcomes between subjects in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | NA [NA to NA] — Only 1 of 17 subjects was referred for or completed spirometry testing (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of spirometric COPD subjects in practices and potential correlation of outcomes between individuals in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster. | 0 [NA to NA] — 0% (0 out of 8 participants) were referred to a specialist for respiratory evaluation/treatment. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits.

97. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 7.6 [1.9 to 13.3] | 8.7 [2.8 to 14.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.80, Generalized estimating equation contrast; Difference in proportion = -1.1, 95% CI 2-sided [-9.3 to 7.1] — [estimate comment as in outcome 1, analysis 1]

98. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 Who Are Referred for or Complete Pulmonary Rehabilitation
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program. | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program.

99. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 Who Are Referred for or Complete Pulmonary Rehabilitation
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 4.5 [0.8 to 8.2] | 8.4 [4.0 to 12.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.18, Generalized estimating equation contrast; Difference in proportion = -3.9, 95% CI 2-sided [-9.7 to 1.8] — [estimate comment as in outcome 1, analysis 1]

100. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled Before March 20, 2019 Who Receive a Recommendation for or Administration of Influenza Vaccination
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 88
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 17 | 8
percent | 88.25 [73.23 to 103.27] | 88.42 [67.34 to 109.51]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.99, Generalized estimating equation contrast; Difference in proportion = -0.17, 95% CI 2-sided [-26.06 to 25.72] — [estimate comment as in outcome 1, analysis 1]

101. Secondary Outcome: Proportion of Participants With Spirometric COPD Enrolled on or After March 20, 2019 Who Receive a Recommendation for or Administration of Influenza Vaccination
Description: as for outcome 28
Time Frame: Baseline to 12 months
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 109 | 111
percent | 87.5 [80.6 to 94.4] | 90.1 [83.7 to 96.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.59, Generalized estimating equation contrast; Difference in proportion = -2.6, 95% CI 2-sided [-12.0 to 6.8] — [estimate comment as in outcome 1, analysis 1]

102. Secondary Outcome: Proportion of Mild COPD Participants Enrolled Before 3/20/2019 With Any of :1) Clinical Spirometry Referral, 2) New COPD Diagnosis, 3) Newly Prescribed Respiratory Medication, 4) Respiratory Specialist Referral, 5) Referral/Completion of Pulmonary Rehab
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory
  Mild COPD = post-bronch FEV1/FVC<0.7 plus 1) FEV1 ≥ 60% and 2) No prior COPD exacerbation
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) aren't based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome
  EUC proportion = intercept. Intervention proportion = intercept + slope Intervention - EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcome between subjects in same practice
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for mild COPD enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — 0% (0 out of 10 participants) met the components of the primary endpoint. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits. | NA [NA to NA] — Only 2 out of 7 subjects were referred for or completed spirometry testing (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of spirometric COPD subjects in practices and potential correlation of outcomes between subjects in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster.

103. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 Who Meet Any of the Components of the Primary Endpoint
Description: Proportion of participants with mild COPD enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Mild COPD is defined as participants with abnormal spirometry, defined as post-bronchodilator FEV1/FVC<0.7 plus both of the following: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
Time Frame: Baseline to 12 months
Population: Only participants that met the criteria for mild COPD enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 30.8 [17.9 to 43.7] | 28.9 [18.7 to 39.1]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.82, Generalized estimating equation contrast; Difference in proportion = 1.9, 95% CI 2-sided [-14.5 to 18.4] — [estimate comment as in outcome 1, analysis 1]

104. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 Referred for or Completion of Clinical Spirometry Testing (Abbreviated as Proportion in the Description)
Description: Mild COPD = post-bronch FEV1/FVC<0.7 plus: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are on the scale from 0% to 100%. Ie. 50.0 = 50% met outcome.
  EUC proportion = intercept. Intervention proportion = intercept + slope.
  Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference).
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcomes between subjects in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 102
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — 0% of participants in this analysis were referred for or competition of spirometry testing. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits. | 0 [NA to NA] — 0% of participants in this analysis were referred for or competition of spirometry testing. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits.

105. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 20.1 [10.3 to 29.9] | 12.5 [6.2 to 18.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney); Difference in proportion = 7.6, 95% CI 2-sided [-4.1 to 19.3] — [estimate comment as in outcome 1, analysis 1]

106. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 With a New Diagnosis of COPD (Abbreviated as Proportion in the Description)
Description: Mild COPD = post-bronchodilator FEV1/FVC<0.7 plus: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome
  EUC proportion = intercept. Intervention proportion = intercept + slope. Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and correlation of outcomes between subjects in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 102
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — 0% of participants in this analysis received a new diagnosis of COPD In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits. | NA [NA to NA] — Only 1 subject was referred for or completed spirometry testing (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of spirometric COPD subjects in practices and potential correlation of outcomes between individuals in the same practice and aren't reported. In general, raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster.

107. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 With a New Diagnosis of COPD
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 12.8 [4.3 to 21.3] | 7.9 [1.9 to 13.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.36, Generalized estimating equation contrast; Difference in proportion = 4.9, 95% CI 2-sided [-5.5 to 15.3] — [estimate comment as in outcome 1, analysis 1]

108. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 With a Newly Prescribed Respiratory Medication (Abbreviated as Proportion in the Description)
Description: Respiratory medication = long acting bronchodilator or anti-inflammatory for respiratory condition.
  Mild COPD = post-bronchodilator FEV1/FVC<0.7 plus: 1) FEV1 ≥ 60% and 2) No prior history of exacerbation of COPD
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits (CL) are not based on raw data proportions. Reported units are from 0% to 100%. Ie. 50.0 = 50% met outcome
  EUC proportion = intercept. Intervention proportion = intercept + slope. Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for different numbers of subjects in practices and c
Time Frame: Baseline to 12 months
Population: as for outcome 102
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — 0% (0 out of 10 participants) received referral for or completed of clinical spirometry testing. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits. | NA [NA to NA] — Only 1 out of 7 subjects was referred for or completed spirometry testing (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of spirometric COPD subjects in practices and potential correlation of outcomes between individuals in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster.

109. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 With a Newly Prescribed Respiratory Medication
Description: as for outcome 37
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 19.6 [9.2 to 30.1] | 15.0 [8.2 to 21.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.47, Generalized estimating equation contrast; Difference in proportion = 4.6, 95% CI 2-sided [-7.9 to 17.1] — [estimate comment as in outcome 1, analysis 1]

110. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 102
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — No participants were referred to a respiratory specialist (insufficient for model convergence). | 0 [NA to NA] — No participants were referred to a respiratory specialist (insufficient for model convergence).

111. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 6.7 [0.3 to 13.1] | 6.1 [0.6 to 11.5]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.88, Generalized estimating equation contrast; Difference in proportion = 0.6, 95% CI 2-sided [-7.8 to 9.0] — [estimate comment as in outcome 1, analysis 1]

112. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 102
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program (insufficient for model convergence). | 0 [NA to NA] — No participants were referred for or competition of pulmonary rehabilitation program (insufficient for model convergence).

113. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 4.0 [-0.2 to 8.1] | 8.2 [1.8 to 14.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.27, Generalized estimating equation contrast; Difference in proportion = -4.3, 95% CI 2-sided [-12.0 to 3.4] — [estimate comment as in outcome 1, analysis 1]

114. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled Before March 20, 2019 Who Received a Recommendation or Administration of Influenza Vaccination
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 10 | 7
percent | 77.75 [49.80 to 105.70] | 82.7 [50.04 to 115.35]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.82, Generalized estimating equation contrast; Difference in proportion = -4.94, 95% CI 2-sided [-47.92 to 38.04] — [estimate comment as in outcome 1, analysis 1]

115. Secondary Outcome: Proportion of Participants With Mild COPD Enrolled on or After March 20, 2019 Who Received a Recommendation or Administration of Influenza Vaccination
Description: as for outcome 35
Time Frame: Baseline to 12 months
Population: as for outcome 103
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 76 | 73
percent | 86.3 [77.7 to 94.9] | 87.4 [77.2 to 97.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.87, Generalized estimating equation contrast; Difference in proportion = -1.1, 95% CI 2-sided [-14.5 to 12.2] — [estimate comment as in outcome 1, analysis 1]

116. Secondary Outcome: Proportion of Participants With Preserved Ration, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with preserved ration, impaired spirometry (PRISm) enrolled before March 18, 2020 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISM enrolled before March 20, 2019 were analyzed for this measure.
  Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | 29.03 [15.4 to 42.6] | 66.7 [35.3 to 98.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.03, Generalized estimating equation contrast; Difference in proportion = -37.6, 95% CI 2-sided [-71.8 to -3.5] — [estimate comment as in outcome 1, analysis 1]

117. Secondary Outcome: Proportion of Participants With Preserved Ration, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with preserved ration, impaired spirometry (PRISm) enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Preserved ratio, impaired spirometry (PRISm) is defined as participants without spirometrically defined COPD who have post-bronchodilator FEV1 < 80% predicted.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 31.2 [25.7 to 36.6] | 28.8 [23.1 to 34.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.56, Generalized estimating equation contrast; Difference in proportion = 2.3, 95% CI 2-sided [-5.6 to 10.3] — [estimate comment as in outcome 1, analysis 1]

118. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | 18.21 [17.49 to 18.93] | 41.27 [16.95 to 65.60]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.06, Generalized estimating equation contrast; Difference in proportion = -23.07, 95% CI 2-sided [-47.40 to 1.27] — [estimate comment as in outcome 1, analysis 1]

119. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 17.6 [12.6 to 22.7] | 14.4 [9.3 to 19.6]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.39, Generalized estimating equation contrast; Difference in proportion = 3.2, 95% CI 2-sided [-4.0 to 10.4] — [estimate comment as in outcome 1, analysis 1]

120. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 With New Diagnosis of COPD
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | 7.33 [1.99 to 12.67] | 9.05 [-6.59 to 24.68]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.84, Generalized estimating equation contrast; Difference in proportion = -1.72, 95% CI 2-sided [-18.24 to 14.80] — [estimate comment as in outcome 1, analysis 1]

121. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 With New Diagnosis of COPD
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 7.5 [4.0 to 11.1] | 5.5 [2.2 to 8.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.42, Generalized estimating equation contrast; Difference in proportion = 2.0, 95% CI 2-sided [-2.9 to 6.9] — [estimate comment as in outcome 1, analysis 1]

122. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 With a Newly Prescribed Respiratory Medication
Description: as for outcome 44
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | 13.17 [4.04 to 22.31] | 55.27 [24.42 to 86.12]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.01, Generalized estimating equation contrast; Difference in proportion = -42.09, 95% CI 2-sided [-74.27 to -9.92] — [estimate comment as in outcome 1, analysis 1]

123. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 With a Newly Prescribed Respiratory Medication
Description: as for outcome 44
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 18.3 [13.3 to 23.2] | 15.8 [11.4 to 20.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.47, Generalized estimating equation contrast; Difference in proportion = 2.4, 95% CI 2-sided [-4.2 to 9.1] — [estimate comment as in outcome 1, analysis 1]

124. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | 17.60 [10.39 to 24.81] | 29.87 [5.46 to 54.27]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.34, Generalized estimating equation contrast; Difference in proportion = -12.27, 95% CI 2-sided [-37.72 to 13.18] — [estimate comment as in outcome 1, analysis 1]

125. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 12.6 [8.4 to 16.7] | 10.2 [6.6 to 13.7]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.39, Generalized estimating equation contrast; Difference in proportion = 2.4, 95% CI 2-sided [-3.1 to 7.9] — [estimate comment as in outcome 1, analysis 1]

126. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | NA [NA to NA] — Only 4 participants were referred for competition of pulmonary rehabilitation program (insufficient for model convergence) in the Intervention Arm. | 0 [NA to NA] — No participants were referred for competition of pulmonary rehabilitation program (insufficient for model convergence) in the Enhanced Usual Care Arm.

127. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 3.5 [0.8 to 6.3] | 4.7 [1.4 to 8.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.59, Generalized estimating equation contrast; Difference in proportion = -1.2, 95% CI 2-sided [-5.5 to 3.1] — [estimate comment as in outcome 1, analysis 1]

128. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled Before March 20, 2019 Who Receive a Recommendation for or Administration of Influenza Vaccination (Abbreviated as Proportion in the Description)
Description: Preserved ratio, impaired spirometry (PRISm) = participants without spirometrically defined COPD who have post-bronch FEV1 < 80% predicted.
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits are not based on raw data proportions. Reported units are on the scale from 0% to 100%. Ie. 50.0 = 50% met outcome.
  EUC proportion = intercept. Intervention proportion = intercept + slope.
  Intervention minus EUC proportion = slope. Ie. 10.0 = Intervention met outcome 10% more than EUC (absolute difference).
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for the different numbers of subjects in practices and correlation of outcomes in the same practice.
Time Frame: Baseline to 12 months
Population: as for outcome 116
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 45 | 9
percent | NA [NA to NA] — Only 5 of 45 subjects didn't receive a recommendation for the vaccine (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of vaccine administration in practices and potential correlation of outcomes between individuals in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster. | 100 [NA to NA] — 100% (9 out of 9 participants) received recommendations for or administration of influenza vaccine. In this case, the raw number of 100% is reported without corresponding (unavailable) confidence limits.

129. Secondary Outcome: Proportion of Participants With Preserved Ratio, Impaired Spirometry (PRISm) Enrolled on or After March 20, 2019 Who Receive a Recommendation for or Administration of Influenza Vaccination
Description: as for outcome 42
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for PRISm enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 226 | 180
percent | 84.7 [79.2 to 90.1] | 84.3 [77.8 to 90.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.94, Generalized estimating equation contrast; Difference in proportion = 0.3, 95% CI 2-sided [-8.2 to 8.8] — [estimate comment as in outcome 1, analysis 1]

130. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with symptomatic non-obstructed (SNO) enrolled before March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC < 0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10. The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled before March 20, 2019 were analyzed for this measure. Participants enrolled before March 20, 2019 completed their 1 year follow-up prior to the COVID-19 pandemic onset.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 35.8 [23.1 to 48.4] | 35.2 [33.2 to 37.1]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.93, Generalized estimating equation contrast; Difference in proportion = 0.6, 95% CI 2-sided [-12.2 to 13.4] — [estimate comment as in outcome 1, analysis 1]

131. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Who Meet Any of the Components of the Primary Endpoint.
Description: Proportion of participants with symptomatic non-obstructed (SNO) enrolled on or after March 20, 2019 who meet one of the following (composite endpoint): 1) referral for clinical spirometry testing, 2) new diagnosis of COPD, 3) newly prescribed respiratory medication (long acting bronchodilator or anti-inflammatory for respiratory condition), 4) referral to a specialist for respiratory evaluation/treatment, or 5) referral for or completion of pulmonary rehabilitation.
  Symptomatic non-obstructed (SNO) is defined as participants without spirometrically defined COPD (post-bronchodilator FEV1/FVC < 0.7) and without PRISm (post-bronchodilator FEV1 ≥ 80% predicted) who have a COPD Assessment Test score ≥ 10. The COPD Assessment Test (CAT) is an 8-item questionnaire that measures the impact of COPD on a person's life. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 25.5 [16.2 to 34.9] | 33.7 [23.5 to 43.9]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.25, Generalized estimating equation contrast; Difference in proportion = -8.2, 95% CI 2-sided [-22.0 to 5.7] — [estimate comment as in outcome 1, analysis 1]

132. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 21.7 [13.1 to 30.4] | 25.1 [21.7 to 28.5]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.48, Generalized estimating equation contrast; Difference in proportion = -3.4, 95% CI 2-sided [-12.7 to 6.0] — [estimate comment as in outcome 1, analysis 1]

133. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Referred for or Completion of Clinical Spirometry Testing
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 17.1 [9.6 to 24.5] | 13.1 [6.1 to 20.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.45, Generalized estimating equation contrast; Difference in proportion = 3.9, 95% CI 2-sided [-6.3 to 14.2] — [estimate comment as in outcome 1, analysis 1]

134. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 With a New Diagnosis of COPD (Abbreviated as Proportion in the Description)
Description: SNO = post-bronch FEV1/FVC ≥ 0.7 and post-bronch FEV1 ≥ 80% predicted and a COPD Assessment Test (CAT) score ≥ 10. The CAT is scored 0-40. Higher score = more severe COPD
  The generalized estimating equation (GEE) model for the Proportion:
  Proportion = intercept (Enhanced Usual Care (EUC) parameter) + slope (Intervention vs. EUC difference). Exchangeable correlation within practice assumed. GEE proportion estimates and confidence limits not based on raw data proportions. Reported units are on the scale from 0% - 100%. Ie. 50 = 50% met outcome
  EUC proportion = intercept. Intervention proportion = intercept + slope
  Intervention - EUC proportion = slope. Ie 10 = Intervention met outcome 10% > EUC (absolute difference)
  When the GEE model does not converge, raw numbers other than 0% or 100% are inappropriate to report, CL are unavailable. Raw proportions do not account for the different numbers of subjects in practices and correlation of outcomes in the same practice
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | NA [NA to NA] — Only 4 of 74 participants received a new diagnosis of COPD (insufficient for GEE model convergence). Raw proportions don't sufficiently account for different numbers of new COPD diagnoses in practices, and potential correlation of outcomes between individuals in the same practice and aren't reported. Raw proportions and corresponding GEE based model estimates for these proportions aren't equivalent in cluster randomized trials with different sample sizes in each cluster. | 0 [NA to NA] — 0% (0 of 20 participants) received a new diagnosis of COPD. In this case, the raw number of 0% is reported without corresponding (unavailable) confidence limits.

135. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 With a New Diagnosis of COPD
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 4.4 [0.2 to 8.7] | 6.7 [2.2 to 11.1]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.48, Generalized estimating equation contrast; Difference in proportion = -2.2, 95% CI 2-sided [-8.4 to 3.9] — [estimate comment as in outcome 1, analysis 1]

136. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Newly Prescribed Respiratory Medication
Description: as for outcome 51
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 14.8 [7.8 to 21.7] | 15.2 [-3.5 to 33.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.97, Generalized estimating equation contrast; Difference in proportion = -0.4, 95% CI 2-sided [-20.4 to 19.5] — [estimate comment as in outcome 1, analysis 1]

137. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Newly Prescribed Respiratory Medication
Description: as for outcome 51
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for symptomatic non-obstructed (SNO) enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 10.6 [3.7 to 17.6] | 22.7 [13.6 to 31.8]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.04, Generalized estimating equation contrast; Difference in proportion = -12.1, 95% CI 2-sided [-23.5 to -0.6] — [estimate comment as in outcome 1, analysis 1]

138. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 8.1 [4.3 to 11.9] | 9.9 [8.5 to 11.2]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.39, Generalized estimating equation contrast; Difference in proportion = -1.8, 95% CI 2-sided [-5.8 to 2.3] — [estimate comment as in outcome 1, analysis 1]

139. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Referred to a Specialist for Respiratory Evaluation/Treatment
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: as for outcome 137
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 4.5 [0.1 to 8.9] | 11.7 [5.5 to 18.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.06, Generalized estimating equation contrast; Difference in proportion = -7.3, 95% CI 2-sided [-14.9 to 0.4] — [estimate comment as in outcome 1, analysis 1]

140. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 4.1 [-0.7 to 8.9] | 5.0 [-1.2 to 11.3]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.82, Generalized estimating equation contrast; Difference in proportion = -0.9, 95% CI 2-sided [-8.8 to 7.0] — [estimate comment as in outcome 1, analysis 1]

141. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Referred for or Completion of Pulmonary Rehabilitation
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 6.2 [0.8 to 11.6] | 5.6 [0.7 to 10.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.86, Generalized estimating equation contrast; Difference in proportion = 0.6, 95% CI 2-sided [-6.6 to 7.9] — [estimate comment as in outcome 1, analysis 1]

142. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled Before March 20, 2019 Who Receive a Recommendation or Administration of Influenza Vaccination.
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: as for outcome 130
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 74 | 20
percent | 87.4 [79.6 to 95.1] | 94.8 [88.6 to 101.0]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.14, Generalized estimating equation contrast; Difference in proportion = -7.4, 95% CI 2-sided [-17.3 to 2.5] — [estimate comment as in outcome 1, analysis 1]

143. Secondary Outcome: Proportion of Participants With Symptomatic Non-obstructed (SNO) Enrolled on or After March 20, 2019 Who Receive a Recommendation or Administration of Influenza Vaccination.
Description: as for outcome 49
Time Frame: Baseline to 12 months
Population: Only participants who met the criteria for SNO enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 112 | 107
percent | 77.0 [68.6 to 85.4] | 88.2 [81.7 to 94.8]

144. Secondary Outcome: Proportion of CAPTURE+ Participants Currently Smoking at Baseline Who Received Over-the-counter Patches/Gum for Smoking Cessation
Time Frame: Baseline to 12 months
Population: Only Capture positive participants currently smoking at baseline who had follow-up data available for over-the-counter patches/gum cessation programs were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 49 | 25
percent | 41.52 [28.48 to 54.57] | 56.18 [37.39 to 74.98]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.21, Generalized estimating equation contrast; Difference in proportion = -14.66, 95% CI 2-sided [-37.54 to 8.22] — [estimate comment as in outcome 1, analysis 1]

145. Secondary Outcome: Proportion of CAPTURE+ Participants Who Experience Hospitalizations
Description: as for outcome 2
Time Frame: Baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 226 | 161
Participants
  Hospitalized for respiratory illness during follow-up | 4 | 2
  No hospitalized for respiratory illness during follow-up | 221 | 158
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care: COPD Education; Test type: Superiority; p = 0.76, Generalized estimating equation contrast; Difference in proportion = 0.4, 95% CI 2-sided [-2.0 to 2.7]

146. Secondary Outcome: Number of Enrolled CAPTURE+ Participants Who Experience Mortality
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Analysis population is CAPTURE positive participants selected for follow-up. This analysis population does not require a follow-up survey to be completed, hence the size of this analysis population differs from analyses requiring a follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care: COPD Education
Number analyzed (Participants) | 331 | 225
Participants | 2 | 2

147. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Experience Hospitalizations
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 46 | 13
percent | 0.0 [NA to NA] — No patients were hospitalized for respiratory illnesses (insufficient variability for confidence limits). | 0.0 [NA to NA] — No patients were hospitalized for respiratory illnesses (insufficient variability for confidence limits).

148. Secondary Outcome: Proportion of CAPTURE+ Participants Enrolled on or After March 20, 2019 Who Experience Hospitalizations
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Only CAPTURE+ participants enrolled on or after March 20, 2019 were analyzed for this measure.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 180 | 148
percent | 2.1 [0.1 to 4.2] | 1.5 [-0.3 to 3.4]
Statistical Analysis 1: Comparison: Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results vs Enhanced Usual Care Arm: COPD Education; Test type: Superiority; p = 0.66, Generalized estimating equation contrast; Difference in proportion = 0.6, 95% CI 2-sided [-2.1 to 3.4] — [estimate comment as in outcome 1, analysis 1]

149. Secondary Outcome: Number of CAPTURE+ Participants Enrolled Before March 20, 2019 Who Experience Mortality.
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Analysis population is CAPTURE positive participants selected for follow-up and enrolled prior to March 20, 2019. This analysis population does not require a follow-up survey to be completed, hence the size of this analysis population differs from analyses requiring a follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 72 | 20
Participants | 0 | 0

150. Secondary Outcome: Number of CAPTURE+ Participants Enrolled After March 20, 2019 Who Experience Mortality.
Description: as for outcome 2
Time Frame: Baseline to 12 months
Population: Analysis population is CAPTURE positive participants selected for follow-up and enrolled after March 20, 2019. This analysis population does not require a follow-up survey to be completed, hence the size of this analysis population differs from analyses requiring a follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
Number analyzed (Participants) | 259 | 205
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse events (AE)s occurring at the Baseline Visit only were collected for all participants, per study protocol. Mortality data was only collected via medical records from Baseline to 12 months in individuals identified as CAPTURE+ at baseline. Note that, in contrast, the primary analysis population required completion of the 12-month follow-up survey, which required them to be alive at 12 months.
Description: Adverse events (AE)s occurring at the Baseline Visit only were collected for all participants, per study protocol. Mortality data was only collected via medical records from Baseline to 12 months in individuals identified as CAPTURE+ at baseline. Note that, in contrast, the primary analysis population required completion of the 12-month follow-up survey, which required them to be alive at 12 months.
Arm/Group | Intervention: COPD Education Plus CAPTURE Education and Patient-level CAPTURE Screening Results | Enhanced Usual Care Arm: COPD Education
All-Cause Mortality (participants affected / at risk) | 2/331 | 2/225
Serious Adverse Events (participants affected / at risk) | 0/1118 | 0/886
Other Adverse Events (participants affected / at risk) | 0/1118 | 0/886

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03583099/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03583099/SAP_001.pdf